CLINICAL TRIAL: NCT00644800
Title: An Open, Multicenter, Non-Comparative Study To Assess The Efficacy And Tolerability Of Intramuscular Ziprasidone Followed By Oral Ziprasidone In Patients With Acute Psychosis
Brief Title: A Study of the Efficacy and Safety of Intramuscular Ziprasidone Followed by Oral Ziprasidone for the Treatment of Psychosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281074
Record Dates: First submitted 2008-03-20; First posted 2008-03-27 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia; Mania; Delusional Disorder; Acute Exacerbation of Psychosis
MeSH Terms: conditions — Schizophrenia; Mania; Schizophrenia, Paranoid | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental)
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — Intramuscular ziprasidone 10 or 20 mg at the investigator's discretion for 1 to 3 days followed by oral ziprasidone capsules 40 to 80 mg twice daily at the investigator's discretion to complete 7 days of treatment
  Other Names: Geodon, Zeldox

SUMMARY:
To assess the efficacy, safety, and tolerability of intramuscular ziprasidone in the treatment of the acute exacerbation of non-organic psychosis of any etiology, including schizophrenia, acute mania, delusional disorder and others.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with psychosis
* Eligible for intramuscular treatment
* Miminum score of 60 on the PANSS, a score of 14 in the sum of PANSS excitation score and a score of at least 4 in 1 of the following items: poor control of impulses, tension, hostility, uncooperativeness or excitation.

Exclusion Criteria:

* Treatment with antidepressants or mood stabilizers within seven days prior to the enrollment; for monoamine oxidase inhibitors (MAOIs) and moclobemide, this period must be two weeks; for fluoxetine, five weeks
* Resistance to conventional antipsychotic agents
* A history of epilepsy
* A diagnosis of abuse of substance within the previous 3 months according to the DSMIV criteria.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2003-07; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale (PANSS) excitation items scores | Days 1-3 (end of intramuscular dosing)

SECONDARY OUTCOMES:
Electrocardiogram at Visits 1 and 5 | Visits 1 (Screening) and 5 (Day 7)
Adverse events at Visits 2, 3, 4, and 5 | Visits 2 (Day 1), 3 (Day 1, 2, 3, or 4), 4 (Day 5), and 5 (Day 7)
Change from baseline in Patient Preference Scale (PPS) scores at Visits 3 and 5 | Visits 2 (Day 1), 3 (Day 1, 2, 3, or 4) and 5 (Day 7)
Laboratory tests at Visits 1 and 5 | Visits 1 (Screening) and 5 (Day 7)
Movement disorder rating scale scores (Barnes Akathisia Scale and Extrapyramidal Symptoms Rating Scale) at Visits 2, 3, 4, and 5 | Visits 2 (Day 1), 3 (Day 1, 2, 3, or 4), 4 (Day 5), and 5 (Day 7)
Change from baseline in PANSS excitation items scores at Visits 3, 4, and 5 | Visits 1 (Screening), 2 (Day 1), 3 (Day 1, 2, 3, or 4), 4 (Day 5), and 5 (Day 7)
Blood pressure and pulse at Visits 1, 2, and 5 | Visits 1 (Screening), 2 (Day 1), and 5 (Day 7)
Change from baseline in Clinical Global Impression-Severity (CGI-S) scores at Visits 3, 4, and 5 | Visits 1 (Screening), 2 (Day 1), 3 (Day 1, 2, 3, or 4), 4 (Day 5), and 5 (Day 7)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Brazil (8):
  - Pfizer Investigational Site, Fortaleza, Ceará
  - Pfizer Investigational Site, Salvador, Estado de Bahia
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, São Gonçalo, Rio de Janeiro
  - Pfizer Investigational Site, Jardim Santa Monica SN, Salvador - BA
  - Pfizer Investigational Site, São Paulo, São Paulo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281074&StudyName=A%20study%20of%20the%20efficacy%20and%20safety%20of%20intramuscular%20ziprasidone%20followed%20by%20oral%20ziprasidone%20for%20the%20treatment%20of%20psychosis